CLINICAL TRIAL: NCT00005061
Title: A Phase I, Open Label Multiple Dose, Safety and Pharmacokinetic Study of Intravenously Administered Humanized Anti-VEGF Monoclonal Antibody (HuMV833) to Patients With Relapsed or Refractory Solid Tumors
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-13992; EORTC-13992; PDL-833-601
Record Dates: First submitted 2000-04-06; First posted 2004-04-12 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bevacizumab

INTERVENTIONS:
Biological: bevacizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the preliminary tolerability and safety of monoclonal antibody VEGF (MOAB VEGF) in patients with relapsed or refractory progressive solid tumors. II. Determine the optimum biologically active dose of MOAB VEGF for further evaluation based on exploratory methods. III. Determine the maximum tolerated dose of MOAB VEGF in these patients. IV. Determine a safe dose of MOAB VEGF for further clinical studies. V. Determine the dose limiting toxicity and pharmacokinetics of this regimen in these patients. VI. Determine the response rate in patients treated with this regimen.

OUTLINE: This is a dose escalation, multicenter study. Patients receive monoclonal antibody VEGF (MOAB VEGF) IV over 1 hour on days 1, 15, 22, and 29. Patients with partial response (PR), complete response (CR), or stable disease (SD) after completion of the fourth dose may receive weekly infusions for up to 6 months in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of MOAB VEGF until the maximum tolerated dose (MTD) and optimum biologically active dose (OBAD) are determined. The MTD is defined as the dose at which 1 of 6 patients experiences dose limiting toxicity. The OBAD is defined as the dose at which vascular endothelial growth factor is optimally inhibited. Patients with PR, CR, or SD are evaluated every 6 weeks until disease progression or initiation of another treatment. Patients who discontinue treatment prematurely due to toxicity are followed weekly until resolution of any associated toxicity. Patients who discontinue treatment after the fourth dose of MOAB VEGF for any reason other than toxicity are followed every month for up to 6 months.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven relapsed or refractory progressive solid tumor that is not amenable to treatment with standard therapies No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Postmenopausal Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL No bleeding or clotting abnormalities Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST or ALT no greater than 2.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: Normal cardiac function by 12 lead ECG Other: No unstable systemic disease or uncontrolled infection that would preclude study participation No concurrent infection requiring antibiotics Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 70 days after study No psychologic, familial, sociologic, or geographic condition that could preclude compliance HIV negative HTLV-1 negative Hepatitis B surface antigen negative No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix No allergy to protein therapeutics

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: At least 4 weeks since prior hormonal antitumor therapy No concurrent steroids or hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Concurrent radiotherapy allowed Surgery: Greater than 4 weeks since prior surgery except biopsy or fine needle aspiration of tumor masses Other: At least 4 weeks since other prior investigational drugs or therapies No other concurrent anticancer treatments No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1999-12; Primary Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, MD, Study Chair — The Christie NHS Foundation Trust
Locations (4):
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Academisch Ziekenhuis Utrecht, Utrecht
- University Hospital of Linkoping, Linköping, Sweden
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom